CLINICAL TRIAL: NCT01484964
Title: A Phase I, Single-Dose, Open-Label, Three-Period, Randomized, Crossover Study to Compare the Relative Bioavailability Between Two Tablet Formulations of ASP015K and to Assess the Food Effect on a New Formulation in Healthy Volunteers
Brief Title: A Single Oral Dose Study to Compare the Bioavailability Between Two Different Tablet Formulations and Assess if There is a Food Effect With the New Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 015K-CL-PK19
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Pharmacokinetics of ASP015K; Bioavailability of ASP015K; Healthy Subjects
Keywords: ASP015K; healthy subjects; bioavailability; food effect; rheumatoid arthritis; psoriasis; transplantation
MeSH Terms: conditions — Arthritis, Rheumatoid; Psoriasis | interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): ASP015K Formulation 1 with moderate-fat meal
  Interventions: Drug: ASP015K
- Treatment B (Experimental): ASP015K Formulation 2 under fasting conditions
  Interventions: Drug: ASP015K
- Treatment C (Experimental): ASP015K Formulation 2 with moderate-fat meal
  Interventions: Drug: ASP015K

INTERVENTIONS:
Drug: ASP015K — oral

SUMMARY:
The purpose of this study is to determine the bioavailability and pharmacokinetics between two different formulations of ASP015K tablets and determine the food effect on the absorption of the new formulation.

DETAILED DESCRIPTION:
Eligible subjects will be admitted on Day -2 and remain confined on the unit for 20 days. Each subject will receive a single dose of study drug per the defined treatment periods on the morning of Day 1, Day 8 and Day 15. There will be a minimum of 7 days between each consecutive dose group.

For Treatment A, Formulation 1 tablets will be administered within 30 minutes after the start of a standard FDA moderate-fat breakfast. Treatment B, Formulation 2 tablets will be administered in a fasted state. For Treatment C, Formulation 2 tablets will be administered within 30 minutes after the start of a standard FDA moderate-fat breakfast.

Any subject discontinuing the study prior to completion should have all end of study evaluations completed

ELIGIBILITY:
Inclusion Criteria:

* Subject weighs at least 45 kg and has a body mass index (BMI) of 18-32 kg/m2
* Male subject agrees to sexual abstinence, is surgically sterile or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method until 90 days after the last dose of study drug administration
* Male subject agrees to not donate sperm until 90 days after the dose of study drug administration
* Female subject is surgically sterile or is post-menopausal and is not pregnant and is not lactating
* Subject's 12-lead electrocardiogram (ECG) is normal
* Subject must be capable of swallowing multiple tablets
* Subject is willing to take and complete the moderate-fat breakfast within 30 minutes

Exclusion Criteria:

* Subject has a previous history of any clinically significant gastro-intestinal, neurological, renal, hepatic, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease, malignancy excluding non-melanoma skin cancer or any other medical condition
* Subject has had major GI surgery (such as colectomy, cholecystectomy, etc)
* Subject has a history of consuming more than 14 units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/ substance abuse within past 2 years
* Subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week
* Subject has a positive test for hepatitis C antibody, or positive test for hepatitis B surface antigen (HBsAg), or positive hepatitis B core antibody
* Subject has a history of the human immunodeficiency virus (HIV) antibody
* Subject has a positive tuberculosis (TB) skin test, Quantiferon Gold test or T-SPOT® test
* Subject received any vaccine within 60 days
* Subject received an experimental agent within 30 days
* Subject has an absolute neutrophil count (ANC) < 2500 cells/mm3
* Subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days
* Subject has a history of smoking or has used tobacco-containing products and nicotine or nicotine-containing products in the past six months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic parameters of ASP015K: C max, AUClast, and AUCinf | Up to Day 18

SECONDARY OUTCOMES:
Composite of pharmacokinetic parameters of ASP015K: tmax, apparent terminal elimination half-life (t1/2), apparent body clearance after oral dosing (CL/F), and apparent volume of distribution (Vz/F) | Up to Day 18
Composite of pharmacokinetic parameters of ASP015K metabolite H2: Cmax, AUClast, AUCinf, tmax and t1/2 | Up to Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development
Locations (1):
- PAREXEL, Glendale, California, United States